CLINICAL TRIAL: NCT02147626
Title: Heart Health 4 Moms: Engaging Women With a Recent History of Preeclampsia to Reduce Their Cardiovascular Disease Risk
Brief Title: Heart Health 4 Moms Trial to Reduce CVD Risk After Preeclampsia
Acronym: HH4M
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Preeclampsia Foundation (Other)
Responsible Party: Principal Investigator, Janet Rich-Edwards, Associate Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2014P002765; CER-1306-02603 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2014-05-20; First posted 2014-05-28 (Estimated); Results first posted 2021-02-15 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-01

CONDITIONS: Cardiovascular Disease; Preeclampsia; Hypertension; Post-partum Weight Retention
Keywords: preeclampsia; cardiovascular disease; health behaviors; behavioral intervention; web-based; Hypertension; Post-partum Weight Retention
MeSH Terms: conditions — Cardiovascular Diseases; Pre-Eclampsia; Hypertension; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Information and Screening Group (Active Comparator): Intervention: The patient website will include the American Heart Association (AHA) Class I Lifestyle recommendations (translated to an 8th grade reading level and with a link to the publication), a link to the online National Institutes of Health (NIH) Dietary Approaches to Stop Hypertension (DASH) website, and the NIH smoking cessation website
  Interventions: Behavioral: Information and Screening Group
- HH4M Intervention Arm (Experimental): Intervention: The HH4M patient website will include information and tools. These resources are customized to help new mothers achieve the AHA Class I Lifestyle recommendations for women with a history of preeclampsia.
  Interventions: Behavioral: Web-based educational and motivational modules; Behavioral: Information and Screening Group

INTERVENTIONS:
Behavioral: Web-based educational and motivational modules
  Arms: HH4M Intervention Arm
Behavioral: Information and Screening Group

SUMMARY:
This study will compare two arms in a randomized clinical trial of cardiovascular risk prevention in women with a history of preeclampsia. The first arm will provide postpartum patients and their clinicians with the American Heart Association's (AHA) Class I Lifestyle Recommendations for women with a history of preeclampsia. The second arm will additionally receive access to a customized patient-informed online program with modules on how to achieve the AHA recommendations for diet, activity and weight management.

DETAILED DESCRIPTION:
The study team will work with patients via focus groups to develop a novel internet-based program to provide information and tools for cardiovascular disease (CVD) risk reduction for women who are at increased risk of CVD by virtue of their history of preeclampsia, a common complication of pregnancy. The American Heart Association has recently issued guidelines that physicians should include history of the hypertensive pregnancy disorder, preeclampsia, as a risk factor for CVD. Indeed, research demonstrates that roughly 2 out of 3 women with a history of preeclampsia will die from CVD. This study will work with patients with prior preeclampsia and with the Preeclampsia Foundation, a patient- based organization, to create an online lifestyle modification program ( accessible by computer or smart phone) for women with recent preeclampsia to reduce CVD risk. The study is a randomized controlled trial to test the program's acceptability, use, and impact on diet, postpartum weight retention, physical activity, blood pressure, and patient knowledge and self-efficacy to improve health.

ELIGIBILITY:
Inclusion Criteria:

* Within 5 years of a live birth complicated by preeclampsia as determined by medical chart review
* Age >=18
* Not pregnant
* Normotensive or prehypertensive
* Access to the internet via computer or mobile device
* Able to communicate in English or Spanish at an 8th grade level.

Exclusion Criteria:

* Type 1 or Type 2 diabetes
* Currently pregnant
* Diagnosis of hypertension BP >140/90 mm Hg or on medications for treatment of hypertension

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 151 (Actual)
Dates: Start 2015-09-21 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet Rich-Edwards, ScD, Principal Investigator — Brigham and Women's Hospital; Ellen Seely, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital;, Boston, Massachusetts, United States

REFERENCES:
- [Background] Sallis JF, Grossman RM, Pinski RB, Patterson TL, Nader PR. The development of scales to measure social support for diet and exercise behaviors. Prev Med. 1987 Nov;16(6):825-36. doi: 10.1016/0091-7435(87)90022-3. PMID 3432232
- [Background] Chasan-Taber L, Schmidt MD, Roberts DE, Hosmer D, Markenson G, Freedson PS. Development and validation of a Pregnancy Physical Activity Questionnaire. Med Sci Sports Exerc. 2004 Oct;36(10):1750-60. doi: 10.1249/01.mss.0000142303.49306.0d. PMID 15595297
- [Background] Mosca L, Ferris A, Fabunmi R, Robertson RM; American Heart Association. Tracking women's awareness of heart disease: an American Heart Association national study. Circulation. 2004 Feb 10;109(5):573-9. doi: 10.1161/01.CIR.0000115222.69428.C9. Epub 2004 Feb 4. PMID 14761901
- [Background] Kim C, McEwen LN, Piette JD, Goewey J, Ferrara A, Walker EA. Risk perception for diabetes among women with histories of gestational diabetes mellitus. Diabetes Care. 2007 Sep;30(9):2281-6. doi: 10.2337/dc07-0618. Epub 2007 Jun 15. PMID 17575087
- [Background] Apovian CM, Murphy MC, Cullum-Dugan D, Lin PH, Gilbert KM, Coffman G, Jenkins M, Bakun P, Tucker KL, Moore TJ. Validation of a web-based dietary questionnaire designed for the DASH (dietary approaches to stop hypertension) diet: the DASH online questionnaire. Public Health Nutr. 2010 May;13(5):615-22. doi: 10.1017/S1368980009991996. Epub 2009 Nov 16. PMID 19912673
- [Result] Rich-Edwards JW, Stuart JJ, Skurnik G, Roche AT, Tsigas E, Fitzmaurice GM, Wilkins-Haug LE, Levkoff SE, Seely EW. Randomized Trial to Reduce Cardiovascular Risk in Women with Recent Preeclampsia. J Womens Health (Larchmt). 2019 Nov;28(11):1493-1504. doi: 10.1089/jwh.2018.7523. Epub 2019 Jun 19. PMID 31215837

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From July 2015 to May 2016, women living in the United States with recent preeclampsia were recruited through the website and social media of the Preeclampsia Foundation, the March of Dimes Foundation, BabyCenter.com, and Craigslist.
Pre-assignment Details: Women were eligible to participate if they had preeclampsia in the past five years and did not have current chronic hypertension; women also had to have access to the internet via computer or mobile device
Groups:
- Information and Screening Group: Intervention: The patient website will include the American Heart Association (AHA) Class I Lifestyle recommendations (translated to an 8th grade reading level and with a link to the publication), a link to the online National Institutes of Health (NIH) Dietary Approaches to Stop Hypertension (DASH) website, and the NIH smoking cessation website
  Information and Screening Group
- HH4M Intervention Arm: Intervention: The HH4M patient website will include information and tools. These resources are customized to help new mothers achieve the American Heart Association ( AHA) Class I Lifestyle recommendations for women with a history of preeclampsia.
  Web-based educational and motivational modules
  Information and Screening Group
Period: Overall Study
Arm/Group | Information and Screening Group | HH4M Intervention Arm
Started | 75 | 76
Completed | 70 | 69
Not Completed | 5 | 7
Not completed — Lost to Follow-up | 4 | 4
Not completed — Pregnancy | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Women with a history of preeclampsia within the past five years were recruited via social media from the United States
Groups:
- Information and Screening Group: Intervention: The patient website will include the AHA Class I Lifestyle recommendations (translated to an 8th grade reading level and with a link to the publication), a link to the online National Institutes of Health (NIH) DASH website, and the NIH smoking cessation website
  Information and Screening Group
- HH4M Intervention Arm: Intervention: The HH4M patient website will include information and tools. These resources are customized to help new mothers achieve the AHA Class I Lifestyle recommendations for women with a history of preeclampsia.
  Web-based educational and motivational modules
  Information and Screening Group
- Total: Total of all reporting groups
Arm/Group | Information and Screening Group | HH4M Intervention Arm | Total
Number analyzed (Participants) | 75 | 76 | 151
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 75 | 76 | 151
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 76 | 151
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Non-Hispanic White | 63 | 61 | 124
  Race/Ethnicity: Non-Hispanic African-American | 2 | 2 | 4
  Race/Ethnicity: Non-Hispanic Asian | 1 | 2 | 3
  Race/Ethnicity: Non-Hispanic Multi-race | 2 | 1 | 3
  Race/Ethnicity: Hispanic/Latina | 7 | 10 | 17
Personal Health Self-efficacy (Eating) [Mean (Standard Deviation); unit: units on a scale] | 4.3 (0.6) | 4.4 (0.6) | 4.4 (0.6)
Personal Health Self-efficacy (Physical Activity) [Mean (Standard Deviation); unit: units on a scale] | 3.9 (0.8) | 3.9 (0.7) | 3.9 (0.7)
Physical Activity [Mean (Standard Deviation); unit: METS/week] | 26.3 (20.1) | 23.5 (16.8) | 24.9 (18.5)
Physical inactivity [Mean (Standard Deviation); unit: hours/week] | 24.4 (14.9) | 22.7 (15.3) | 23.5 (15.1)
Adherence to Dietary Approaches to Stop Hypertension (DASH) Diet [Mean (Standard Deviation); unit: units on a scale] | 23.1 (4.8) | 24.4 (4.9) | 24.3 (5.1)
Patient Knowledge of Cardiovascular Disease Risk [Mean (Standard Deviation); unit: units on a scale] | 2.0 (0.9) | 1.9 (0.8) | 2.0 (0.8)
Patient Control Over Cardiovascular Disease Risk [Mean (Standard Deviation); unit: units on a scale] | 3.2 (0.4) | 3.2 (0.4) | 3.2 (0.4)

OUTCOME MEASURES:

1. Primary Outcome: Eating Habits Confidence Survey
Description: The Eating Habits Confidence Survey measures the self-efficacy of a patient to improve their diet. Scores range from 1 (low self-efficacy) to 5 (high self-efficacy). A higher score is a better outcome.
Time Frame: 9 months after intervention starts
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Information and Screening Group | HH4M Intervention Arm
Number analyzed (Participants) | 70 | 69
units on a scale | 4.2 (0.7) | 4.5 (0.6)

2. Primary Outcome: Exercise Confidence Survey
Description: The Exercise Confidence Survey measures self-efficacy of patient to increase physical activity Scores range from 1 (low self-efficacy) to 5 (high self-efficacy). A higher score is a better outcome.
Time Frame: 9 months after intervention starts
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Information and Screening Group | HH4M Intervention Arm
Number analyzed (Participants) | 70 | 69
units on a scale | 3.7 (1) | 4 (0.7)

3. Primary Outcome: DASH Online Questionnaire
Description: The DASH Online Questionnaire is a food frequency questionnaire that prompts recall of daily servings of foods and beverages consumed in the past 30 days. We calculate a DASH score based on daily intake of eight components (fruits, vegetables, nuts and legumes, whole grains, low-fat dairy, sodium, lean meats and poultry, and sweets). Quintile rankings were summed across components to obtain a summary DASH score for each participant that ranged from 8 to 40. A higher score indicates higher DASH compliance.
Time Frame: 9 months after intervention starts
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Information and Screening Group | HH4M Intervention Arm
Number analyzed (Participants) | 70 | 69
units on a scale | 23.6 (4.8) | 24.5 (4.7)

4. Primary Outcome: Pregnancy Physical Activity Questionnaire
Description: The Pregnancy Physical Activity Questionnaire is a validated questionnaire for women that includes activities relevant to caring for young children. Our measure ascertained type, duration, and frequency of recreational activity and childcare activity. It also measured inactivity (sedentary behavior), such as reading, using a computer, and watching television. The time spent in each activity is multiplied by its intensity measured in Metabolic Equivalent of Task Value (METS) to yield the average weekly energy expenditure related to that activity. The score ranged from 0 to 113 METS per week.
Time Frame: 9 months after intervention starts
Measure: Mean (Standard Deviation); unit: METs/week
Arm/Group | Information and Screening Group | HH4M Intervention Arm
Number analyzed (Participants) | 70 | 69
METs/week | 25.8 (18.2) | 26.6 (19.5)

5. Primary Outcome: Physical Inactivity in the Pregnancy Physical Activity Questionnaire
Description: The Pregnancy Physical Activity Questionnaire is a validated questionnaire for women that includes activities relevant to caring for young children. Our measure ascertained type, duration, and frequency of recreational activity and childcare activity. It also measured inactivity (sedentary behavior), such as reading, using a computer, and watching TV. The time spent in each inactivity was summed. The hours per week of reported inactivity ranged from 0 to 85.
Time Frame: 9 months after intervention starts
Measure: Mean (Standard Deviation); unit: Hours/week
Arm/Group | Information and Screening Group | HH4M Intervention Arm
Number analyzed (Participants) | 70 | 69
Hours/week | 22.7 (16.5) | 16.5 (10.7)

6. Primary Outcome: Patient Knowledge of Cardiovascular Disease Risk
Description: Adapted from 2012 American Heart Association National Survey of women's knowledge of their cardiovascular disease (CVD) risk; adaptation is knowledge of risk with respect to preeclampsia history. The score ranges from 1 (low knowledge) to 4 (high knowledge).
Time Frame: 9 months after intervention starts
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Information and Screening Group | HH4M Intervention Arm
Number analyzed (Participants) | 70 | 69
units on a scale | 2.5 (0.9) | 2.7 (0.8)

7. Primary Outcome: Patient Control Over Cardiovascular Disease Risk
Description: To assess women's sense of personal control over their health, we adapted Kim and Walker's survey on perception of chronic diabetes risk among women with a history of gestational diabetes, using factor analysis (with varimax rotation) to reduce seven items from the Kim scales to a single factor we named ''Personal Control over Cardiovascular Disease Risk.'' The resulting measure had a Cronbach's alpha of 0.73. The score ranges from 1 (low control) to 4 (high control). High control is a better outcome.
Time Frame: 9 months after intervention starts
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Information and Screening Group | HH4M Intervention Arm
Number analyzed (Participants) | 70 | 69
units on a scale | 3.2 (0.4) | 3.2 (0.4)

ADVERSE EVENTS:
Time Frame: 9 months after start of intervention
Arm/Group | Information and Screening Group | HH4M Intervention Arm
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/69
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/69
Other Adverse Events (participants affected / at risk) | 0/70 | 0/69

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-05): https://cdn.clinicaltrials.gov/large-docs/26/NCT02147626/Prot_SAP_000.pdf